CLINICAL TRIAL: NCT06310291
Title: A Phase 1, First in Human, Randomized, Placebo-controlled Trial With a Controlled Gluten Challenge to Evaluate Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of VTP-1000 in Adults With Celiac Disease
Brief Title: VTP-1000 in Adults With Celiac Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Barinthus Biotherapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GLU001
Record Dates: First submitted 2024-02-16; First posted 2024-03-15 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Celiac Disease
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Intervention Model Description: The Single Ascending Dose part of the trial contains a placebo controlled randomized 4+2 design, where four participants will receive active IMP and two placebo. The Multiple Ascending Dose is a standard sequential design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Matched Placebo (SAD) (Placebo Comparator): 2 placebo comparators; 1 for each part of the study
  Interventions: Other: Matched Placebo
- VTP-1000 Dose 1 (SAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000
- VTP-1000 Dose 2 (SAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000
- VTP-1000 Dose 3 (SAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000
- Matched Placebo (MAD) (Placebo Comparator): 2 placebo comparators; 1 for each part of the study
  Interventions: Other: Matched Placebo
- VTP-1000 Dose 1 (MAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000
- VTP-1000 Dose 2 (MAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000
- VTP-1000 Dose 3 (MAD) (Experimental): 3 dose levels in SAD and MAD parts of trial
  Interventions: Biological: VTP-1000

INTERVENTIONS:
Biological: VTP-1000 — Intramuscular (IM) injection comprised of self-assembling nanoparticles of gluten peptides and a rapamycin component
  Arms: VTP-1000 Dose 1 (MAD); VTP-1000 Dose 1 (SAD); VTP-1000 Dose 2 (MAD); VTP-1000 Dose 2 (SAD); VTP-1000 Dose 3 (MAD); VTP-1000 Dose 3 (SAD)
Other: Matched Placebo — Intramuscular (IM) injection comprised of saline solution
  Arms: Matched Placebo (MAD); Matched Placebo (SAD)

SUMMARY:
GLU001 is a first-in-human clinical trial to assess the safety and tolerability of VTP-1000 for adults with celiac disease. This trial will assess VTP-1000 at various dose levels compared to placebo in a single ascending dose (SAD) and multiple ascending dose (MAD) format. Participants will be followed for a short period of time to assess the impact of VTP-1000 on their immune system (Adverse events, reactions in the blood, and physical exam differences). Participants enrolled in the MAD portion of the trial will undergo a gluten challenge to assess the impact exposure to gluten has on participants after administration of VTP-1000.

DETAILED DESCRIPTION:
VTP-1000 is a gluten-derived (GLU) peptide immunotherapy that is designed to induce antigen-specific immune tolerance against gluten in patients with celiac disease. The technology underlying VTP-1000 consists of the sponsor's proprietary self-assembling nanoparticles based on amphiphilic peptides tolerance immunotherapy (SNAP-TI) platform which has been configured to package 12 GLU peptide antigens and rapamycin into nanoparticles of ~20 nm diameter.

The goal of treatment with VTP-1000 is to induce tolerance to gluten in patients with coeliac disease by activating antigen-specific regulatory T (Treg) cells that promote tolerance and reducing pre-existing, pathogenic antigen-specific effector T (Teff) cells that underly disease pathogenesis. In turn, this may allow for better management of the condition.

GLU001 is a multi-center phase I first in human study to assess the safety and tolerability of VTP-1000 in adults with celiac disease. The trial also aims to demonstrate proof-of-principle of induction of immune tolerance and early proof-of-concept for VTP-1000 as a potential treatment for coeliac disease based on assessment of pharmacodynamics and preliminary efficacy determined by means of a controlled gluten challenge.

GLU001 will be conducted as a randomized double-blind placebo-controlled study in two parts - Part A and Part B. Part A will be a single ascending dose (SAD) followed by Part B a multiple ascending dose (MAD) which incorporates a gluten challenge.

Part A (Single Ascending Dose)

A stepwise single dose escalation of 3 dose levels of VTP-1000 is planned. A total of 6 participants will be treated at each dose level (4 will receive VTP-1000 and 2 will receive matched placebo). A sentinel dosing approach will be followed, with the first 2 participants randomized to receive VTP1000 or placebo in a 1:1 ratio. Subsequent participants will be randomized in a 3:1 ratio at least 7 days after the second sentinel participant has received trial intervention. Participants will be screened for eligibility up to 28 days prior treatment. Participants will be followed for 21 days after dosing including a 3-day domicile period following administration of VTP-1000.

Part B (Multiple Ascending Dose)

A stepwise multiple dose escalation of up to 3 dose levels of VTP-1000 is planned. A total of 8 participants will be treated at each dose level (6 will receive VTP-1000 and 2 will receive matched placebo). A sentinel dosing approach will be followed, with the first 2 participants randomized to receive VTP1000 or placebo in a 1:1 ratio. Subsequent participants will be randomized in a 3:1 ratio at least 7 days after the second sentinel participant has received trial intervention. Participants will be screened for eligibility up to 28 days prior to the start of treatment. Eligible participants will receive 3 doses of trial intervention every 2 weeks at a given dose level with and followed for 57 days. After completion of the third dose of trial intervention, participants will undergo a gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease as confirmed by positive serology and intestinal histology
* Presence of Human Leukocyte Antigen (HLA)-DQ2.5 genotype
* Participants who are on a well controlled gluten restricted diet
* Negative or weak positive anti-tissue transglutaminase (tTG) IgA antibodies and negative or weak positive anti-deamidated gliadin peptide IgG (anti-DGP)-IgA/IgA antibodies
* Non-pregnant or breast feeding females
* No other clinical significant findings at screening

Exclusion Criteria:

* Refractory celiac disease
* Selective IgA deficiency
* Positive for HLA-DQ8
* Known wheat allergy or that is Type I hypersensitivity
* Active inflammatory bowel disease or other condition with symptoms that will be similar to celiac disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events, Serious Adverse Events and Adverse Events of Special Interest (AESIs) | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Incidence and severity of treatment-emergent adverse events (TEAEs) , Serious Adverse Events (SAEs) , Adverse Events of Special Interest (AESIs) and adverse events leading to trial intervention discontinuation or trial withdrawal according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities in standard Clinical Chemistry laboratory safety parameters | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Changes from baseline and clinically significant abnormalities in standard clinical laboratory safety parameters according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities in standard Coagulation laboratory safety parameters | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Measurement of in standard clinical laboratory safety parameters according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities in standard hematology laboratory safety parameters | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Measurement of standard hematology clinical laboratory safety parameters according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities in standard urinalysis laboratory safety parameters | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Measurement of standard urinalysis clinical laboratory safety parameters according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities 12-lead electrocardiogram (ECG) parameters | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Changes from baseline and clinically significant abnormalities in 12-lead ECG parameters recorded according to NCI CTCAE Version 5.0
Changes from baseline and clinically significant abnormalities in vital signs | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Changes from baseline and clinically significant abnormalities in vital signs according to NCI CTCAE Version 5.0
Number of participants with changes from baseline in anti-tissue transglutaminase (anti-tTG) immunoglobulin A (IgA) antibodies | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Measurement of anti tTG immunoglobulin at screening and post treatment
Changes in physical examination findings | Participants will be assessed for up to 21 days and 57 days post first dose for SAD and MAD parts of the study respectively.
  Full physical examination required at screening; symptom-directed physical examination at all other clinic visits. Each physical examination must include a review of the administration sites.

SECONDARY OUTCOMES:
PART A SAD:Maximum concentration in plasma (Cmax) rapamycin component | SAD Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
PART A SAD: Time corresponding to Cmax (Tmax) of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
AUC from time 0 to last quantifiable concentration (AUC0-t) of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
AUC extrapolated to infinity (AUC0-∞)of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
Half-life of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
Clearance of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
Volume of distribution of rapamycin component | Day 1 pre-dose; 0.083 hours* (±2 minutes), 0.25 hours* (±5 minutes), 0.5 hours (±5 minutes), 1 hour (±5 minutes), 2 hours (±5 minutes), 4 hours (±10 minutes), 8 hours (±10 minutes), 24 hours (±30 minutes), 48 hours (±2 hours), 120 hours (±3 hours).
  Blood concentration of the rapamycin component of VTP1000 at specified timepoints measured using a liquid chromatography tandem mass spectrometry (LC-MS/MS) method and standard pharmacokinetic parameters
Part B MAD:Maximum concentration in plasma (Cmax) rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The Maximum concentration in plasma (Cmax) results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.
Part B MAD:Time corresponding to Cmax (Tmax) of rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The Cmax(Tmax) results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.
Part B MAD:AUC from time 0 to last quantifiable concentration (AUC0-t) of rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The AUC from time 0 to last quantifiable concentration (AUC0-t) results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.
Part B MAD:AUC extrapolated to infinity (AUC0-∞)of rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The pharmacokinetic results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.
Part B MAD: Half-life of rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The Half-life results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.
Part B MAD: Clearance of rapamycin component | Part B (MAD): Days 1, 15 and 29 pre-dose and 4 hours (±10 minutes) post-dose; Day 43 pre-challenge and Day 50
  The clearance of rapamycin component results will be reviewed from Part A (SAD) and the Part B (MAD) schedule may be updated accordingly to include additional sampling timepoints and inclusion of the derivation of pharmacokinetic parameters, as applicable.

OTHER OUTCOMES:
Gluten Antigen-specific T Cell Responses - Enzyme linked immunospot (ELISpot) | Part A (SAD): Day 1 pre-dose, Days 8 and 15 Part B (MAD): Day 1 pre-dose, Days 8, 22 and 36, Day 43 pre-challenge, Days 50 and 57
  Peripheral Blood Mononucleocytes (PBMCs) will be isolated at the trial site or at a Central Laboratory. Following PBMC isolation, analysis of the magnitude of gluten antigen-specific T cell responses (Treg and Teff) in peripheral blood will be performed by the sponsor using enzyme linked immunospot (ELISpot)
T cell receptor (TCR) sequencing | Part A (SAD): Day 1 pre-dose, Day 15 Part B (MAD): Day 1 pre-dose, Day 43 pre-challenge and Day 57
  Whole Blood sampling with sequencing The whole blood will be isolated, frozen and stored at -80°C until shipped for analysis. Full details on blood sample collection, processing and handling requirements will be provided in the Laboratory Manual
Serum Cytokine Concentrations | SAD Day 1 pre-dose, 4 hours and 24 hours postdose MAD: Days 1, 15 and 29 pre-dose and 4 hours post-dose
  2 mL whole blood samples will be drawn for evaluation of Interleukin 2 (IL-2) in serum.Samples will be stored at -80°C until shipped to a Central Laboratory for analysis. Full details on blood sample collection, processing and handling requirements will be provided in the Laboratory Manual.
  Analysis of IL-2 concentration (and optionally additional cytokines) will be performed at the Central Laboratory using a multiplex cytokine (Meso Scale Discovery S-plex) method as specified in the respective Analytical Protocol.
Cytokine Whole Blood Stimulation | Part A (SAD): Day 1 pre-dose, Days 8 and 15 Part B (MAD): Day 1 pre-dose, Days 8, 22 and 36, Day 43 pre-challenge and Days 50 and 57
  Five 4 mL samples will be drawn and transferred to Greiner Item Number 454088 Vacuette® tubes containing stimulation cocktails for evaluation of cytokines in whole blood stimulated with GLU peptide antigens.Samples will be incubated for 24 hours before processing to sera and stored at -80°C until shipped for analysis. Full details on blood sample collection, processing and handling requirements will be provided in the Laboratory Manual.
  Analysis of sera will be performed at a Central Laboratory using a single or multiplex cytokine method as specified in the respective Analytical Protocol.

CONTACTS AND LOCATIONS:
Locations (16):
- United States (16):
  - Parexel EPCU LA, Los Angeles, California
  - Peak Gastroenterology Associates, Colorado Springs, Colorado
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - GCP Research, St. Petersburg, Florida
  - Parexel EPCU Baltimore, Baltimore, Maryland
  - Clinical Research Institute of Michigan, Clinton Township, Michigan
  - West Michigan Clinical Research Center, Wyoming, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone - Gastroenterology Associates, New York, New York
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Centricity Research, Columbus, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - PPD Research Unit, Austin, Texas
  - Velocity Clinical Research, Salt Lake City, West Jordan, Utah
  - Clinical Research Partners, Richmond, Virginia
  - Velocity Clinical Research, Seattle, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No